CLINICAL TRIAL: NCT04993261
Title: Evaluation of Dual Energy CT for the Detection of Gastrointestinal Carcinoids
Brief Title: An Investigational Scan (Dual Energy CT) in Detecting Gastrointestinal Carcinoid Tumors
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-0578; NCI-2019-02477 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0578 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-07-21; First posted 2021-08-06 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Carcinoid Syndrome; Carcinoid Tumor; Digestive System Neuroendocrine Tumor G1; Metastatic Carcinoid Tumor
MeSH Terms: conditions — Serotonin Syndrome; Carcinoid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (dual energy CT scan) (Experimental): Patients undergo one dual energy CT scan during scheduled CT scan.
  Interventions: Procedure: Dual-Energy Computed Tomography

INTERVENTIONS:
Procedure: Dual-Energy Computed Tomography — Undergo dual energy CT scan
  Other Names: DECT

SUMMARY:
This trial studies the use of a special type of computed (CT) scan called dual energy CT in detecting gastrointestinal carcinoid tumors. CT is an imaging technique that uses x-rays and a computer to create images of areas inside the body. Dual energy computed tomography is a technique used during routine CT scans to help obtain and process the image after the scan is complete. Doctors want to learn if dual energy computed tomography can help improve the detection of carcinoid tumors during routine CT scans.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate prospectively the sensitivity and specificity of dual energy computed tomography (CT) in detecting primary gastrointestinal (GI) carcinoid.

OUTLINE:

Patients undergo one dual energy CT scan during scheduled CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Patients with: clinical features of carcinoid syndrome (or) increased serum and urinary markers suggestive of carcinoid (or) endoscopic biopsy proven carcinoid (or) metastases which are biopsy proven as carcinoid.
* Patient is scheduled to have a clinically indicated staging CT exam.
* Patients who have signed their informed consent form to undergo the study.

Exclusion Criteria:

* Patients who have already had their primary GI carcinoid resected.
* Contraindication to intravenous contrast agents (e.g. allergy, renal failure, dialysis, pregnancy etc.).
* Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2015-09-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of dual energy computed tomography in detecting primary gastrointestinal carcinoid tumors | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ajaykumar Morani, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States